CLINICAL TRIAL: NCT06751342
Title: Using Psychophysics Methods to Investigate Sensory Dominance After Cataract Surgery
Status: Active, not recruiting | Type: Observational
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Yune Zhao, Vice president of Eye Hospital of Wenzhou Medical University, Wenzhou Medical University
Other Study IDs: psychophysical methods
Record Dates: First submitted 2024-12-20; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- Subjects with Unilateral Congenital Cataract Undergoing Surgery
- Subjects with Bilateral Congenital Cataract Undergoing Surgery
- Control Group of Children
- Subjects with Comparable Degrees of Bilateral Age-Related Cataract
- Subjects with Different Degrees of Bilateral Age-Related Cataracts
- Subjects with Shallow Anterior Chambers in Both Eyes

SUMMARY:
Using Psychophysics Methods for Quantitative Assessment of Sensory Binocular Imbalance After Cataract Surgery

DETAILED DESCRIPTION:
Using binocular phase combination paradigms and binocular rivalry paradigms to quantitatively assess the degree of sensory binocular imbalance in patients following cataract surgery, investigating the relationship between unilateral and bilateral cataracts in children and varying severities of cataracts in adults with respect to sensory ocular dominance, and forecasting the postoperative quality of life for patients.

ELIGIBILITY:
Inclusion Criteria:

1. Ages between 6 and 90 years old, and the individual or legal guardian is capable of understanding and voluntarily signing an informed consent form;
2. No history of ocular trauma or intraocular surgery, no physical or medical treatments have been undergone, and the clinical diagnosis in the medical records is age-related, congenital, or developmental cataract patients;
3. Best-corrected visual acuity in both eyes is greater than 0.8 before the study, fusion ability is normal as checked by Worth's 4-dot test, and at least 1 month has passed since the last surgery;
4. Good communication skills and the ability to understand and grasp the trial;
5. No significant contraindications to surgery found in preoperative systemic and ocular examinations.

Exclusion Criteria:

1. Patients with traumatic or complex cataracts;
2. Those diagnosed with glaucoma before or after surgery;
3. Individuals with a history of intraocular surgery (such as vitrectomy) or laser treatment;
4. Exclude those with severe ocular comorbidities (including microphthalmia, aphakia, anterior segment dysgenesis, uveitis, optic nerve dysplasia, retinopathy of prematurity, congenital glaucoma, etc.) and severe systemic comorbidities (including syndromes affecting connective tissue function, such as Marfan syndrome, homocystinuria, or Down syndrome, severe birth defects, and epilepsy);
5. Any systemic diseases related to the eyes, such as rheumatic immune diseases;
6. Those with surgical records indicating any severe intraoperative complications during cataract surgery;
7. Individuals who cannot cooperate with the examination.

Ages: 6 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Included in Eye Hospital of Wenzhou Medical University for "phacoemulsification combined with intraocular lens implantation"
Sampling Method: Probability Sample
Enrollment: 96 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Perceptual Phase | Each subject undergoes a one-time examination, which lasts for about a year. Each subject's participation in this clinical study will take approximately 0.5 hour.
  The perceptual phase when the interocular contrast between the two eyes is 1.
Ocular Dominance Index (ODI) | Each subject undergoes a one-time examination, which lasts for about a year. Each subject's participation in this clinical study will take approximately 0.5 hour.
  The ratio of the total time spent by the observer reporting complete dominance of visual stimuli presented to the dominant or non-dominant eye.

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthalmology and Optometry Hospital, Wenzhou, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No